CLINICAL TRIAL: NCT01892085
Title: Adequate Breast Milk for Improved Health of Very Low Birth Weight Preterm Infants
Brief Title: Early Initiation of Milk Expression in Mothers of Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-00071-N; 1R15NR013566-01A1 (NIH); IRB201200071 (Other: Univeristy of Florida)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Breast Milk Expression
Keywords: Breast milk; lactogenesis stage two; premature infant; insufficient milk supply; breast milk expression
MeSH Terms: conditions — Breast Milk Expression; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early initiation (Experimental): Initiation of breast milk expression <1 hour following delivery.
  Interventions: Behavioral: Early initiation
- Intermediate expression (Experimental): Initiation of milk expression 1-<3 hours following delivery.
  Interventions: Behavioral: Intermediate expression
- Late initiation (Other): Initiation of milk expression >3-6 hours following delivery.
  Interventions: Behavioral: Late initiation

INTERVENTIONS:
Behavioral: Early initiation — Initiation of breast milk expression <1 hour following delivery.
  Other Names: Early initiation of breast milk expressed
  Arms: Early initiation
Behavioral: Intermediate expression — Initiation of milk expression 1-<3 hours following delivery.
  Other Names: Intermediate timing of breast milk expression
  Arms: Intermediate expression
Behavioral: Late initiation — Initiation of milk expression >3-6 hours following delivery.
  Other Names: Late initiation of breast milk expression.
  Arms: Late initiation

SUMMARY:
Compelling evidence exists that breast milk helps protect very premature infants from prematurity-specific morbidities. Unfortunately, mothers of premature infants often exhibit delayed lactogenesis stage II (when the milk "comes in") and decreased breast milk production. Several studies have linked earlier initiation of breast milk expression following delivery with a greater milk production. However, none conclusively determined the optimal timing of breast milk expression. As a result these mothers continue to struggle with inadequate breast milk production. This study will follow 180 mothers of premature infants for 6 weeks following delivery to test

Earlier initiation of breast milk expression following delivery is associated with (1) an earlier lactogenesis stage II, (2) greater volume of breast milk production during the first 6 weeks, (3) improved short-term infant health outcomes and (4) women who deliver at an earlier gestation will have decreased milk production and a later lactogenesis stage II. Following stratification according to the gestational age of the infant (23-27 weeks vs. 28-32 weeks), eligible women will be randomly assigned to one of three groups and instructed to start mechanically expressing their r breasts, either in the first hour, 1-3 hours or 3-6 hours following delivery. The timing of lactogenesis stage II will be documented, and the volume of breast milk produced will continue to be measured for the first 6 weeks following delivery and at discharge. Infant nutritional outcomes will be measured throughout the 6-week study. The impact of the differences in timing of initiation of milk expression following delivery on timing of lactogenesis stage II, milk volume, short term nutritional outcomes, amount of breast milk feedings at discharge, and impact of gestational age on milk volume and lactogenesis stage II will be determined.

DETAILED DESCRIPTION:
Mothers will be randomly assigned to one of three groups. Group 1 will begin pumping their breasts with the assistance of medical or nursing personnel within 60 minutes following delivery. Group 2 will begin pumping their breasts with the assistance of medical or nursing personnel within 1- less than 3 hours following delivery. Group 3 will begin pumping their breasts with the assistance of medical or nursing personnel 3-6 hours following delivery. Mothers will also do the following

1. Complete a log with information about their daily breast pumping sessions for 6 weeks.
2. Bring your breast milk to the neonatal intensive care unit when they visit and the milk will be weighed to determine the volume of milk.
3. Episodes of kangaroo care (placing the infant on your bare chest) will be collected.
4. Receive a call beginning the day after you delivery and then daily until their milk comes in to ask about a feeling of fullness in their breasts.

In addition the following will be done

1. If their infant breastfeeds, he/she will be weighed before and after feeding to collect data on how much milk he/she ate from the breast
2. Information regarding infant's weekly breast milk intake and breast milk intake at discharge will be collected

ELIGIBILITY:
Inclusion Criteria:

* 1) at least 18 years of age,
* 2) English or Spanish-speaking,
* 3) stated intent to breastfeed,
* 4) anticipating the birth of a very low birth weight infant (≤1500 grams) between 23-32 weeks gestation.

Exclusion Criteria:

* 1) known illicit maternal drug use,
* 2) history of breast reduction or augmentation,
* 3) positive HIV status,
* 4) mother not transported to recovery by 45 minutes following delivery or
* 5) infant not expected to live over 2 weeks following delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-11; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Parker, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands, Gainesville, Florida, United States

REFERENCES:
- [Derived] Parker LA, Sullivan S, Cacho N, Krueger C, Mueller M. Effect of Postpartum Depo Medroxyprogesterone Acetate on Lactation in Mothers of Very Low-Birth-Weight Infants. Breastfeed Med. 2021 Oct;16(10):835-842. doi: 10.1089/bfm.2020.0336. Epub 2021 Apr 28. PMID 33913765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Started | 58 | 62 | 60
Completed | 52 | 61 | 55
Not Completed | 6 | 1 | 5
Not completed — Death | 4 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation | Total
Number analyzed (Participants) | 52 | 61 | 55 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (5.4) | 26.1 (6.4) | 28.2 (6.1) | 26.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 61 | 55 | 168
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 8 | 18
  Not Hispanic or Latino | 47 | 56 | 47 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 23 | 19 | 65
  White | 21 | 32 | 29 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 7 | 18
Region of Enrollment [Number; unit: participants]
  United States | 52 | 61 | 55 | 168

OUTCOME MEASURES:

1. Primary Outcome: Pumped Milk Volume Day 1
Description: Volume of pumped milk on day 1 postpartum
Time Frame: Day 1 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 3 (3) | 4 (4) | 5 (4)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.015, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.339, Marginalized two part model

2. Primary Outcome: Pumped Milk Volume on Day 2
Description: Volume of breast milk pumped on day 2 postpartum
Time Frame: Day 2 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 11 (11) | 13 (12) | 15 (12)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.024, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.317, Marginalized two part model

3. Primary Outcome: Pumped Milk Volume Day 3
Description: Volume of milk pumped on day 3 postpartum
Time Frame: Day 3 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 31 (30) | 36 (31) | 41 (31)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.031, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.298, Marginalized two part model

4. Primary Outcome: Pumped Milk Volume Day 4
Description: Volume of pumped milk on Day 4 postpartum
Time Frame: Day 4 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 73 (70) | 82 (70) | 94 (72)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.05, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.27, Marginalized 2 part model

5. Primary Outcome: Pumped Milk Volume on Day 5
Description: Volume of pumped milk on Day 5 postpartum
Time Frame: Day 5 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 145 (138) | 157 (135) | 180 (138)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.069, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.244, Marginalized two part model

6. Primary Outcome: Pumped Milk Volume Day 6
Description: Volume of pumped milk on Day 6 postpartum
Time Frame: Day 6 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 60
mL | 240 (230) | 253 (217) | 293 (233)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.094, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.235, Marginalized 2 part model

7. Primary Outcome: Pumped Milk Volume on Day 7
Description: Volume of milk pumped on day 7 postpartum
Time Frame: Day 7 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 337 (322) | 343 (294) | 400 (305)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.123, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.210, Marginalized two part model

8. Primary Outcome: Pumped Milk Volume at Day 14
Description: Volume of pumped milk on day 14 postpartum
Time Frame: Day 14 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 398 (380) | 391 (335) | 461 (352)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.143, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.196, Marginalized two part model

9. Primary Outcome: Pumped Milk Volume Day 21
Description: Volume of milk pumped on day 21 postpartum
Time Frame: Day 21 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 396 (370) | 377 (305) | 447 (341)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.185, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.183, Marginalized two part model

10. Primary Outcome: Pumped Milk Volume Day 28
Description: Volume of milk pumped on day 28 postpartum
Time Frame: Day 28 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 332 (317) | 305 (262) | 365 (275)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.229, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.170, Marginalized two part model

11. Primary Outcome: Pumped Milk Volume on Day 35
Description: Volume of milk pumped on day 35 postpartum
Time Frame: Day 35 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 234 (224) | 209 (179) | 252 (192)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.314, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.162, Marginalized two part model

12. Primary Outcome: Pumped Milk Volume on Day 42
Description: Volume of milk pumped on day 42 postpartum
Time Frame: Day 42 postpartum
Measure: Least Squares Mean (Standard Deviation); unit: mL
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
mL | 139 (133) | 120 (103) | 146 (112)
Statistical Analysis 1: Comparison: Early Initiation vs Late Initiation; Test type: Superiority; p = 0.377, Marginalized two part model
Statistical Analysis 2: Comparison: Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.149, Marginalized two part model

13. Secondary Outcome: Hours From Birth to Onset of Lactogenesis Stage 2
Description: Mothers were asked daily concerning a feeling of fullness in their breasts as a measure of onset of lactogenesis stage 2
Time Frame: Hours from birth to onset of lactogenesis stage 2
Measure: Mean (Standard Deviation); unit: hours from birth
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
hours from birth | 140.5 (144.7) | 94.7 (65) | 109 (98.4)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.08, ANOVA

14. Secondary Outcome: Days Lactated
Description: Days mothers lactated until infant NICU discharge
Time Frame: birth to approximately 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
days | 45.3 (31.8) | 48.7 (28.2) | 48.2 (28.3)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.82, ANOVA

15. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 1
Description: The percentage of feeds consisting of mother's own milk consumed by the participant's infants from day 1-7
Time Frame: Day 1 to 7
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 71.7 (42.1) | 69.2 (43.4) | 81.9 (36.3)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 00.22, Chi-squared

16. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 2 Consumed by Infants
Description: The percentage of feeds consisting of mother's own milk consumed by the participants infants from day 7-14
Time Frame: Day 7-14
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 65.7 (45.1) | 66.7 (44.1) | 70.2 (45.6)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.87, Chi-squared

17. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 3
Description: The percentage of feeds consisting of mother's own milk consumed by the participant's infant from day 14-21
Time Frame: Day 14-21
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 55.7 (48.5) | 59.6 (48.7) | 70.2 (45.1)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.27, Chi-squared

18. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 4
Description: The percentage of feeds consisting of mother's own milk consumed by the participant's infant from day 21-28
Time Frame: Day 21-28
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 57.5 (48) | 62.3 (46.4) | 64.5 (47.7)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.77, Chi-squared

19. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 5
Description: The percentage of feeds consisting of mother's own milk consumed by the participant's infant from day 28-35
Time Frame: Day 28-35
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 51.8 (49) | 54.3 (48.1) | 65.6 (46.5)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.31, Chi-squared

20. Secondary Outcome: Percentage of Feeds Consisting of Mother's Own Milk Week 6
Description: The percentage of feeds consisting of mother's own milk consumed by the participant's infant from day 35-42
Time Frame: Day 35-42
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
percent | 51.1 (48.9) | 53.9 (49.7) | 56 (48.6)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.90, Chi-squared

21. Secondary Outcome: Percentage of Feedings Consisting of Mother's Own Milk at NICU Discharge
Description: The percentage of feedings consisting of mother's own milk consumed by the participant's infant over the 24 hours period prior to NICU discharge among mothers who continued to lactate
Time Frame: 24 hour period prior to NICU discharge
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
Number analyzed (Participants) | 52 | 61 | 55
Percent | 82 (30.8) | 80 (31.2) | 90 (20)
Statistical Analysis 1: Comparison: Early Initiation vs Intermediate Expression vs Late Initiation; Test type: Superiority; p = 0.36, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Early Initiation | Intermediate Expression | Late Initiation
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/61 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/61 | 0/55
Other Adverse Events (participants affected / at risk) | 0/52 | 0/61 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT01892085/Prot_SAP_000.pdf